CLINICAL TRIAL: NCT05377775
Title: Mesh Stents Study in Iliac Complex Lesions Iliac-Mesh Stent Study (IMS-Study)
Brief Title: Mesh Stents Study in ILIAC Complex Lesions (IMS-Study)
Acronym: IMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WarsawMU IMS v.01
Record Dates: First submitted 2022-04-29; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Peripheral Arterial Disease; Iliac Artery Stenosis; Embolus Arterial; Ischemic Leg
Keywords: Iliac artery stenosis; High-risk plague; Mesh stent; Peripheral embolisation; Peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, open-label, single-arm, non-randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conventional Implantation of mesh stent (Experimental): Conventional Implantation of mesh stent in iliac stenosis with high-risk plaques
  Interventions: Device: Iliac Stenting

INTERVENTIONS:
Device: Iliac Stenting — Conventional Implantation of mesh stent in iliac stenosis with high-risk plaques

SUMMARY:
The main objective of the IMS-Study is to evaluate the short and long-term safety and efficacy of mesh stent implantation in patients with stenotic iliac disease with complex plaques or lesions containing thrombotic material.

DETAILED DESCRIPTION:
Iliac artery disease may include complex lesions with a vulnerable plaque and containing thrombotic materials. The treatment of these complex plaques is frequently complicated with local, acute occlusion, dissection and distal embolisation.

Studies with a mesh stent in the carotid region have shown a reduced risk of peripheral embolization. The use of mesh stents in iliac arteries can provide similar benefits. The structure of the stents, sizes, and the release system do not require any changes. The study is to assess the usefulness of mesh stents in preventing peripheral embolisation.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria (principal):

  * Patients older than 18 years, after Vascular Team evaluation, according to local standards, eligible for Iliac artery
  * Written, informed consent to participate
  * Agreement to attend Protocol required (standard) follow up visits and examinations
* Angiographic Inclusion Criteria (principal):

  * De novo iliac stenosis
  * Stenosis eligible for endovascular treatment per Vascular Team evaluation (according to current standards and guidelines)
  * High-risk morphology stenosis with complex/thrombotic lesions (per 1 independent, experienced operator).

Exclusion Criteria:

* General Exclusion Criteria (principal):

  * Life expectancy <1 year (e.g., active neoplastic disease).
  * Chronic kidney disease with creatinine > 3.0 mg/dL.
  * Coagulopathy.
  * Contraindication for decoagulation
  * History of uncontrolled contrast media intolerance
  * Myocardial infarction in 72 hours preceding the stenting procedure (if possible, postponing the procedure)
  * Stroke in 6 weeks preceding the stenting procedure (if possible, postponing the procedure)
  * Pregnancy (positive pregnancy test)
* AngiographicExclusion Criteria (principal):

  * Chronic total occlusion not amenable to re-canalization
  * Stent in the target vessel/lesion
  * Anatomic variants precluding stent implantation
  * Mobile (free-floating) plaque elements in aorta or arteries proximal to the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-10 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MACNE (Major Adverse Cardiac or Neurological Event ) | 48 hours after procedure
  In-hospital MACNE (death, stroke, myocardial infarction, acute limb or target organ ischemia)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Myrcha, Ass.Prof., Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical Universtity of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Randomized trial comparing CGuard™ stent vs. Wallstent™ — https://pubmed.ncbi.nlm.nih.gov/30266356/
- See also: Thirty-Day Results of the Novel CGuard-Covered Stent in Patients Undergoing Carotid Artery Stenting — https://pubmed.ncbi.nlm.nih.gov/33855877/
- See also: CGuard MicroNet-Covered "One-Size-Fits-All" Carotid Stent — https://pubmed.ncbi.nlm.nih.gov/31060430/
- See also: The IRONGUARD 2 Study — https://pubmed.ncbi.nlm.nih.gov/34391704/
- See also: Analysis from the PARADIGM study — https://pubmed.ncbi.nlm.nih.gov/30945420/